CLINICAL TRIAL: NCT04251702
Title: Two Novel Biomarkers for Labor Dystocia: Developing a Physiologic Understanding to Facilitate Precision in Diagnosis and Individualized Management
Brief Title: Biomarkers of Uterine Muscle Physiology
Acronym: BUMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Nova Biomedical (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-0307; F31NR018582-01 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Labor (Obstetrics)--Complications; Labor; Dyscoordinate
Keywords: labor dystocia; cesarean delivery; uterine monitoring
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and Serum will be frozen and biobanked for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Low-Risk Individuals in Labor: Healthy laboring individuals with a Singleton Term fetus in the Vertex position. Patients requiring medical management of diabetes or hypertension will be excluded.

SUMMARY:
This observational study characterizes the relationship between amniotic fluid lactate and uterine electromyography during labor in healthy individuals at term planning a vaginal birth. Additional comparison measures and outcomes measures will be collected and analyzed as exploratory measures.

DETAILED DESCRIPTION:
Elevated amniotic fluid lactate (AFL) and uterine electromyography (EMG) mathematically transformed to calculated the power density spectrum median frequency have been found separately to be associated with labor dystocia and cesarean birth. Similarly, recent research indicates that the cytokine IL-6 may play a critical role in labor onset and potentially labor progression. All three are hypothesized to reflect that uterine fatigue plays a role in the pathophysiology of labor dystocia for some women.

This study aims to characterize the relationship between these three measures to better understand the role of uterine fatigue in labor dystocia and triangulate biomarkers of fatigue that may lead to a better understanding of labor dystocia phenotypes.

In addition to the primary measures, comparison measures will be collected. For AFL comparison, venous whole blood lactate and capillary lactate will be collected and measured using both a point-of-care lactate meter (Stat Strip Lactate Meter, Nova Biomedical) and a table-top blood gas analyzer (Nova Prime). For EMG comparison, routine contraction monitoring data will be collected and compared to the EMG signal. IL-6 will be measured both in blood and amniotic fluid using a novel microsampling protocol. Three visual analog scales on women's experiences of fatigue, anxiety, and pain will also be administered.

Additional data will be collected from the medical record to perform exploratory and hypothesis generating analysis.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age: 18-41 years at the due date
* Term gestation: 37-41 weeks estimated gestational age (EGA)
* Single fetus in a vertex presentation: Pregnancy with only one fetus that is in a head down position with the occiput leading into the pelvis upon admission to the hospital.

Exclusion Criteria:

* Pre-existing or gestational diabetes requiring medical management: The diagnosis of diabetes of any kind requiring management with medications including but not limited to insulin, glyburide, and metformin as indicated in the health record.
* Pre-existing or gestational hypertension or pre-eclampsia requiring medical management: The diagnosis of hypertension of any kind requiring management with medications including but not limited to long-term hypertension management such as methyldopa and short-term or emergency hypertension management such as labetalol or magnesium sulfate as indicated in the health record.
* Suspected fetal anomaly or intrauterine growth restriction: Any diagnosed fetal anomalies or intrauterine growth restriction as indicated in the health record.
* Use of amnioinfusion prior to sample collection: Amnioinfusion, the infusion of fluids into the uterus using an intrauterine catheter may affect AFL concentrations. Any amnioinfusion prior to sample collection will exclude participants from continued participation.
* Fetal distress prior to or during sample collection: Category 3 fetal heart tracing as defined by the National Institute of Child Health and Development22, absent fetal heart rate variability with recurrent late deceleration, recurrent variable decelerations, bradycardia, or sinusoidal rhythm.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women with a Singleton Term fetus in the Vertex position in labor.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Amniotic Fluid Lactate | During active labor (4-10cm) after rupture of membranes
  Amniotic fluid lactate as measured using the handheld StatStrip Lactate Meter (Nova Biomedical). This will be measured once during active labor (6-10cm) after rupture of membranes.
Median power density spectrum of uterine electromyography | 30 minutes after amniotic fluid collection during active labor (4-10cm) after rupture of membranes
  Uterine electromyography measured using the Bloomlife Lovelace EMG monitor
Visual analog scale for fatigue | At the time of amniotic fluid collection
  Participants indicate their level of fatigue on a 100 mm horizontal line anchored by "no fatigue at all" (0) and "the most serious fatigue imaginable" (100). The scale will be administered at the time of amniotic fluid collection.
Amniotic fluid IL-6 | At the time of amniotic fluid collection
  Amniotic fluid collected using a volumetric assisted microsampling device.

SECONDARY OUTCOMES:
Capillary Lactate | At the time of amniotic fluid collection
  Capillary lactate measured using the handheld StatStrip Lactate Meter (Nova Biomedical). This will be measured within 10 minutes of the amniotic fluid lactate measurement.
Serum Lactate | At the time of amniotic fluid collection
  Serum lactate measured using a POC device and analyzed using a laboratory assay
Serum IL-6 | At the time of amniotic fluid collection
  Serum IL-6 measured using a laboratory assay (multiplex)

OTHER OUTCOMES:
(Exploratory) Maternal Age | At the time of delivery
  Maternal age in years
(Exploratory) Maternal BMI | At the time of delivery
  Maternal body mass index (kg2/cm)
(Exploratory) Neonatal Sex | Identified by provider at time of delivery
  Neonatal sex (male/female)
(Exploratory) Neonatal Weight | Measured by provider at time of delivery
  Neonatal weight (g)
(Exploratory) Perinatal Mood Disorders | During the prenatal period
  Presence of perinatal mood disorders as identified by ICD 10 code, history of perinatal mood disorders recorded in the chart, or Edinburgh Postnatal Depression Score > 13
(Exploratory) Length of Latent Labor | Immediately prior to labor
  length of latent labor in hours measured from the time the participant identifies labor onset through the time of active labor onset identified via partograph
(Exploratory) Length of Active Labor | During labor
  length of active labor in hours measured from the time of active labor onset identified by partograph, until birth
(Exploratory) Oxytocin Augmentation | During labor (prior to birth)
  Use of oxytocin (y/n) during labor
(Exploratory) Fetal distress | During labor
  Fetal distress identified as category 3 fetal heart tracing during labor (Y/N)
(Exploratory) Birth Outcome | At the time of birth
  Vaginal birth, cesarean birth, or instrumental vaginal birth
(Exploratory) Postpartum Hemorrhage | Within the first hour after birth
  Presence of postpartum hemorrhage (Y/N) >1000 ml of blood loss
(Exploratory) Estimated Blood Loss | Within the first hour after birth
  Blood loss (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kissler, PhD, Principal Investigator — University of Colorado Anschutz Medical Campus, College of Nursing
Locations (1):
- UCHealth Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing can be arranged by contacting the PI